CLINICAL TRIAL: NCT04639739
Title: Anti-CD19 CAR NK Cell Therapy for Relapsed or Refractory B Cell Non-Hodgkin Lymphoma: a Multi-center, Uncontrolled Trial.
Brief Title: Anti-CD19 CAR NK Cell Therapy for R/R Non-Hodgkin Lymphoma.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Principal Investigator, Xi Zhang, MD, Chef of Hematology Department, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR NK for NHL
Record Dates: First submitted 2020-11-12; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: NHL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19 CAR NK cells (Experimental): The study will employ dose level cohorts of three patients that will be treated at each level described below, based on the number of T cells to be infused using the "3 + 3" dose-escalation strategy to find MTD followed by a dose-expansion phase at determined optimal dosage.
  Interventions: Biological: anti-CD19 CAR NK

INTERVENTIONS:
Biological: anti-CD19 CAR NK — 2×106 /kg、6×106 /kg、2×107/kg Treatment follows a lymphodepletion, the recommended chemotherapy regimen consists of Fludarabine (30 mg/m2 per day) and Cyclophosphamide (500mg/m2 per day) for 3 days prior to cell infusion，the actual regiment is determined by the statue of patients.

SUMMARY:
Although the anti-CD19 CAR-T cell therapies have gained significant results in patients with relapsed and refractory B-cell hematologic malignancies. There are limitations of CAR-T cells, the consuming manufacturing time and expensive price exclude the majority of patients. therefore, we designed this trial to manifest the safety and efficacy of anti-CD19 CAR NK cell therapy in non-Hodgkin lymphoma

ELIGIBILITY:
Subjects must meet the following criteria for inclusion in the study： 1) Male or female subjects between the ages of 18 and 75（including critical values）； 2) Subjects histologically confirmed as diffuse diffuse large B cell lymphoma (DLBCL), transformed follicular lymphoma (TFL), primary mediastinal B cell lymphoma (PMBCL) and mantle cell lymphoma (MCL) ：

1. Refractory B-NHL ：Subjects of which the best response to standard first-line treatment is PD,(those intolerant to first-line treatment will not be included in this study). Subjects of which the best response to at least four courses of first-line treatment is SD, with a duration of SD less than 6 months after the last treatment. Subjects of which the best response to the last course of second-line treatment or above treatments is PD or the best response to at least two courses of second-line treatment or above treatments is SD, with a duration of SD less than 6 months.
2. Relapsed B-NHL：The disease relapses confirmed by histopathology in subjects who achieved complete remission after standard systematic treatment and second-line treatment. Or the disease relapses confirmed by histopathology within 1 year after hematopoietic stem cell transplantation (not limited to the previous therapeutic regimen) ； Male or female subjects between the ages of 18 and 75（including critical values）； Subjects histologically confirmed as diffuse diffuse large B cell lymphoma (DLBCL), transformed follicular lymphoma (TFL), primary mediastinal B cell lymphoma (PMBCL) and mantle cell lymphoma (MCL) ：

Refractory B-NHL ：Subjects of which the best response to standard first-line treatment is PD,(those intolerant to first-line treatment will not be included in this study). Subjects of which the best response to at least four courses of first-line treatment is SD, with a duration of SD less than 6 months after the last treatment. Subjects of which the best response to the last course of second-line treatment or above treatments is PD or the best response to at least two courses of second-line treatment or above treatments is SD, with a duration of SD less than 6 months.

Relapsed B-NHL：The disease relapses confirmed by histopathology in subjects who achieved complete remission after standard systematic treatment and second-line treatment. Or the disease relapses confirmed by histopathology within 1 year after hematopoietic stem cell transplantation (not limited to the previous therapeutic regimen) ；

Subjects with TFL must receive chemotherapy before transformation and meet the above definition of relapse or refractory after transformation.

According to Lugano response criteria 2014, there should be at least one evaluable tumor focus: the longest diameter of intranodal focus > 1.5cm, the longest diameter of extranodal focus > 1.0cm； Positive expression of CD19 in tumor tissue； Subjects who have no effect or relapse after single-target CAR-T treatment can also be included in the group.

Approved anti-tumor therapies, such as systemic chemotherapy, systemic radiotherapy, and immunotherapy, have been completed for at least 2 weeks before the precondition.

ECOG≤1； Life expectancy ≥ 3 months； Neutrophil absolute count ≥ 1×10^9/L； platelet count ≥ 50×10^9/L； Absolute lymphocyte count ≥ 1×10^8/L ；

Adequate organ function reserve :

GPT, GST ≤ 5× UNL（upper normal limit）；

Serum total bilirubin ≤3× UNL； The left ventricular ejection fraction (LVEF) ≥ 50% was diagnosed by echocardiography, and there was no clinically significant pericardial effusion and ECG abnormality； Basic oxygen saturation in indoor natural air environment > 92%； For female subjects of childbearing age, results are negative in urine pregnancy test before screening and administration, and subjects agree to take effective contraceptive measures at least one year after infusion; Male subjects with partners' fertility must agree to use effective barrier contraceptive methods at least one year after infusion, and avoid sperm donation； Voluntary signing of informed consent;

Exclusion Criteria:

Any of the following points shall be deemed as no entry into this study：

Other tumors except cured non-melanoma skin cancer, cervical cancer in situ, superficial bladder cancer, breast duct cancer in situ, or other malignant tumors with complete remission of more than 5 years)；

Severe mental disorders；

A history of genetic diseases such as Fanconi anemia, Shudder-Dale syndrome, Costman syndrome, or any other known bone marrow failure syndrome；

History of allogeneic stem cell transplantation；

Heart disease with grade III-IV heart failure [NYHA classification], myocardial infarction, angioplasty or stenting, unstable angina or other heart diseases with prominent clinical symptoms within one year before admission；

Subjects with any indwelling catheter or drainage tube (such as percutaneous nephrostomy tube, bile drainage tube or pleura/peritoneum/pericardium catheter), should be excluded. (Special central venous catheter is allowed)；

Subjects with a history of CNS lymphoma, CSF malignant cells, or brain metastasis；

Subjects with a history of CNS disease,such as epilepsy, cerebral ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving CNS；

Any of the following virological ELISA results are positive: HIV antibody, HCV antibody, TPPA, HBsAg；

Active infection requiring systematic treatment within 2 weeks before single collection；

Subjects with known severe allergic reactions to cyclophosphamide or fludarabine, or diagnosed as the allergy；

History of autoimmune diseases (e.g. Crohn disease, rheumatoid arthritis, systemic lupus erythematosus) that cause end-organ damage or require systemic immunosuppressive medications or systemic disease modifying drugs in the past 2 years；

Presence of pulmonary fibrosis；

Subjects who have received other clinical trial treatment within 4 weeks before participating in this trial should be excluded. Or the signing date of informed consent is within 5 half-lives of the last application of another clinical trial (whichever is longer)；

Subjects with poor compliance due to physiological, family, social, geographical and other factors, or those unable to cooperate with the study plan or follow-up； At the discretion of the investigator, there are complications requiring systemic corticosteroid therapy (≥ 5mg / day of prednisone or equivalent dose of other corticosteroids) or other immunosuppressive drugs within 6 months after this clinical research treatment；

The lactating woman who is reluctant to stop breastfeeding；

Any other condition considered unsuitable by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2020-12-17 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLTs) | within 4 weeks after infusion
  To characterize the safety, tolerability, and determine the recommended dosage of Anti-CD19 CAR NK Cell Therapy for R/R Non-Hodgkin Lymphoma
Incidence and severity of AEs and SAEs | Up to 24 months
  To characterize the safety, tolerability, and determine the recommended dosage of Anti-CD19 CAR NK Cell Therapy for R/R Non-Hodgkin Lymphoma

SECONDARY OUTCOMES:
The overall response rate(ORR) | 1 and 3 months after infusion
  to characterize the efficacy of Anti-CD19 CAR NK Cell Therapy for R/R Non-Hodgkin Lymphoma
progression-free survival (PFS) | 1, 3, 6, 12 and 24 months after infusion
  to characterize the efficacy of Anti-CD19 CAR NK Cell Therapy for R/R Non-Hodgkin Lymphoma
overall survival(OS) | 1, 3, 6, 12 and 24 months after infusion
  to characterize the efficacy of Anti-CD19 CAR NK Cell Therapy for R/R Non-Hodgkin Lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: Xi Zhang, Study Chair — Xinqiao Hospital of Chongqing
Locations (1):
- Department of Hematology, Xinqiao Hospital, Chongqing, Chongqing Municipality, China